CLINICAL TRIAL: NCT05760222
Title: Early Acupuncture Treatment of Vasomotor Symptoms and Sleep Disorders in Breast Cancer Luteinising Hormone-releasing Hormone Analogues(LHRHa) Induced Menopause: AcuHOTFLASH Study
Brief Title: Acupuncture Treatment of Vasomotor Symptoms in Breast Cancer Patients
Acronym: Acu-HOTFLASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4523
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hot flashes; Acupuncture
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture arm (Experimental): Intervention with 10 acupuncture sessions twice per week for 4 weeks followed by 2 more sessions once per week
  Interventions: Other: Acupuncture
- Usual care arm (No Intervention): Lifestyle recommendations

INTERVENTIONS:
Other: Acupuncture — Acupuncture for prevention/early treatment of vasomotor symptoms and sleep impairment in LHRHa induced amenorrhea in Breast Cancer patients
  Arms: Acupuncture arm

SUMMARY:
The goal of this clinical trial is to evaluate the impact of acupuncture in preventing worsening of hot flashes and sleep disorders in paucisymptomatic premenopausal Breast Cancer (BC) patients undergoing LHRHa plus endocrine therapy.

According to the published data, acupuncture is an effective and long-lasting (6 to 8 months) treatment for severe vasomotor symptoms. Treatment response can be affected by different variables, including intervention timing.

The main question this study aims to answer is:

Can we expect an additional benefit resulting from an early intervention (when patients are still presymptomatic/paucysintomatic) with acupuncture in preventing worsening in terms of frequency/severity of hot flashes and sleep disorders?

Researchers will compare patients randomized in two arms:

Arm A: intervention with acupuncture Arm B: usual care to see if acupuncture is superior to usual care in preventing worsening of hot flashes

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial of superiority of acupuncture compared to usual care for prevention/early treatment of vasomotor symptoms and sleep impairment in LHRHa induced amenorrhea.

The primary endpoint will be a reduction in frequency and intensity of hot flashes in the intervention arm compared to standard care, measured by the Hot Flash Composite Score (HFCS) at 6 months following the protocol. Among the secondary outcomes, sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI) and quality of life by the Menopause-specific Quality of Life Questionnaire (MenQOL) and EORTC Quality of Life Questionnaire (EORTC-C30).

A total of 90 premenopausal BC (stage I-III) patients undergoing LHRHa plus Endocrine Therapy (tamoxifen or aromatase inhibitors) after surgery will be randomized 1:1 in two arms:

Arm A: intervention with 10 acupuncture sessions twice per week for 4 weeks followed by 2 more sessions once per week Arm B: usual care

Participants in both arms will report the hot flash frequency and severity daily (HFCS), and will fill three questionnaires (EORTC QLQ-C30, MenQoL, PSQI) according to the following timeline:

T0 (baseline): 6 weeks following the first LHRHa administration T1: 6 weeks from T0 (corresponding to the end of acupuncture protocol for Arm A) T2: 18 weeks from T0 T3: 30 weeks from T0

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Breast Cancer patients
* Stage I-III breast cancer patients undergoing LHRHa plus ET (tamoxifen or aromatase inhibitors) after surgery
* Informed consent

Exclusion Criteria:

* Ongoing LHRHa during chemotherapy
* Ongoing pharmacological therapy or natural products consumption for vasomotor symptoms
* Metastatic breast cancer
* Ongoing heparin or anticoagulant therapy
* Psychiatric conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Reduction of frequency and intensity of hot flashes following acupuncture treatment | HFCS collected for one week, 6 months following the protocol.
  Hot flashes will be measured by the Hot Flash Composite Score (HFCS)

SECONDARY OUTCOMES:
Sleep quality | PSQI collected 6 months following the protocol.
  Sleep quality will be measured by Pittsburgh Sleep Quality Index (PSQI)
Quality of life (QoL) | MenQOL and EORTC QLQ-C30 will be collected 6 months following the protocol.
  QoL will be measured by Menopause-specific Quality of Life Questionnaire (MenQOL) and EORTC Quality of Life Questionnaire (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Magno, Principal Investigator — Fondazione policlinico Gemelli - IRCCS
Locations (1):
- Fondazione Policlinico Gemelli- IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao JJ, Bowman MA, Xie SX, Bruner D, DeMichele A, Farrar JT. Electroacupuncture Versus Gabapentin for Hot Flashes Among Breast Cancer Survivors: A Randomized Placebo-Controlled Trial. J Clin Oncol. 2015 Nov 1;33(31):3615-20. doi: 10.1200/JCO.2015.60.9412. Epub 2015 Aug 24. PMID 26304905
- [Background] Lesi G, Razzini G, Musti MA, Stivanello E, Petrucci C, Benedetti B, Rondini E, Ligabue MB, Scaltriti L, Botti A, Artioli F, Mancuso P, Cardini F, Pandolfi P. Acupuncture As an Integrative Approach for the Treatment of Hot Flashes in Women With Breast Cancer: A Prospective Multicenter Randomized Controlled Trial (AcCliMaT). J Clin Oncol. 2016 May 20;34(15):1795-802. doi: 10.1200/JCO.2015.63.2893. Epub 2016 Mar 28. PMID 27022113